CLINICAL TRIAL: NCT00251316
Title: The Effects of Lithium Carbonate on Low Dose Radioiodine Ablation in Early Thyroid Cancer Treatment
Brief Title: Effect of Lithium Carbonate on Low-Dose Radioiodine Therapy in Early Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Monica Skarulis, MD, PI, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 060025; 06-DK-0025 (Other: NIH Clinical Center)
Record Dates: First submitted 2005-11-09; First posted 2005-11-09 (Estimated); Results first posted 2012-12-27 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Thyroid Cancer; Differentiated Thyroid Carcinoma
Keywords: Thyroid Neoplasm; I-131; Radiation Dose; Radiation Effect; Pharmaceutical Adjuvant; Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Lithium Carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lithium Carbonate (Experimental): Patients recently diagnosed with papillary or follicular thyroid cancer who have had their thyroid gland removed and whose cancer has not spread beyond the thyroid may be eligible for this study. Participants in this arm receive lithium capsules.
  Interventions: Drug: Lithium Carbonate
- Placebo (Placebo Comparator): Patients recently diagnosed with papillary or follicular thyroid cancer who have had their thyroid gland removed and whose cancer has not spread beyond the thyroid may be eligible for this study. Participants in this arm receive placebo (look-alike capsules with no active ingredient).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lithium Carbonate — 30 mCi of 131I
  Other Names: Lithium carabonate
  Arms: Lithium Carbonate
Drug: Placebo — Patients recently diagnosed with papillary or follicular thyroid cancer who have had their thyroid gland removed and whose cancer has not spread beyond the thyroid may be eligible for this study. Participants in this arm receive placebo (look-alike capsules with no active ingredient).
  Other Names: Identical placebo
  Arms: Placebo

SUMMARY:
This study will examine the safety and effectiveness of using lithium, which has been used to enhance the effectiveness of high-dose 131I, with a single low dose (30 mCi) of 131I for thyroid ablation in patients with recently diagnosed papillary or follicular thyroid cancer who have had their thyroid gland removed and whose cancer has not spread beyond the thyroid.

Participants are randomly assigned to receive lithium capsules or placebo (look-alike capsules with no active ingredient). They follow a low-iodine diet for 2 weeks before starting treatment and are then admitted to the NIH Clinical Center for study and treatment for 11 days, during which they remain on the low-iodine diet. Blood samples are collected almost every day to analyze thyroid hormones, kidney and liver function, lithium concentrations and other tests.

DETAILED DESCRIPTION:
Postsurgical thyroid remnant ablation with (131)I is considered standard clinical care for most cases of papillary and follicular thyroid cancer, to eliminate normal thyroid tissue which may contain microscopic cancer. Furthermore, ablation enhances the sensitivity of subsequent (131)I scanning and serum thyroglobulin (TG) measurement for the detection of recurrent or persistent disease. Low dose (131)I (30 mCi) successfully ablates thyroid remnant in 8-61% of cases. This dose can be repeated and result in overall less radiation exposure than that associated with high dose therapy (100 mCi). Ablation achieved with one or more small doses of radioactive iodine is not associated with decreased survival or cancer recurrence. According to the literature there is no difference in the 30-year recurrence rates between groups receiving low and high dose ablation therapy for well differentiated thyroid cancer without distant metastases at the time of initial therapy. The benefits of using low dose of (131)I are minimization of whole body radiation exposure, reduction in side effects and lower cost. Higher rates of successful ablation by low dose of 131I could be achieved by increasing uptake of (131)I and/or lengthening retention of radioiodine in the remnant thyroid tissue. Recombinant human thyroid-stimulating hormone (rhTSH) has been used successfully to increase radioiodine uptake. Lithium has been used to increase radioiodine retention and has been shown to be useful in the treatment of residual or metastatic cancer. The combination of rhTSH and lithium as adjuncts to 30 mCi radioactive iodine (RAI) ablation therapy in low risk thyroid cancer patients may provide a method that reduces the cumulative dose of radioiodine needed to successfully treat thyroid cancer. The specific aim of this study is to determine whether adjunct lithium carbonate improves the success rate of postsurgical ablation of thyroid remnants using low dose (131)I (30 mCi) and rhTSH in low risk patients with differentiated thyroid carcinoma. Patients with well-differentiated papillary or follicular thyroid cancer stage I or II, according to the National Thyroid Cancer Treatment Cooperative Study (NTCTCS) classification at time of surgery, will be enrolled. Eligible patients will have had a total or near-total thyroidectomy within 6 months of enrollment. This randomized, placebocontrolled, double-blind study will permit an evaluation of the risk/benefit ratio of adding lithium as an adjuvant to the already established method of administering low-dose (131)I ablation therapy, to optimize the (131)I retention. All patients will undergo diagnostic rhTSH (123)I whole body scan at the end of the study to assess the success of thyroid ablation.

ELIGIBILITY:
* INCLUSION CRITERIA

  1. Patients older than 16 years with well-differentiated papillary or follicular thyroid cancer stage I or II, according to the NTCTCS classification at time of surgery
  2. Patients younger than 45 years with any size of primary papillary or follicular tumor
  3. Patients older than 45 years with:

     1. primary papillary tumor less than 4 cm or
     2. primary follicular tumor less than 1 cm
* EXCLUSION CRITERIA

  1. Patients with postsurgical thyroid remnant more than 5 g
  2. Patients with distant metastases
  3. Patients above 45 years of age having:

     1. known cervical lymph nodes metastases
     2. microscopic multifocal follicular cancer
     3. microscopic extraglandular invasion of follicular cancer
     4. gross extraglandular invasion of papillary or follicular cancer
  4. Patients with confirmed histological subtypes of well-differentiated thyroid cancer such as Hurtle cell carcinoma, insular and tall cell variants of papillary cancer.
  5. Pregnant or lactating women
  6. Patients with renal impairment defined as repeat serum creatinine concentrations above 1.5 mg/dl on thyroid hormone
  7. Patients on chronic lithium therapy for psychiatric illness
  8. Patients with current unstable cardiovascular conditions
  9. Patients with severe chronic medical conditions (liver failure, severe debilitation, dehydration, sodium depletion, any other cancer requiring therapy, etc)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica C Skarulis, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Sherman SI. Thyroid carcinoma. Lancet. 2003 Feb 8;361(9356):501-11. doi: 10.1016/s0140-6736(03)12488-9. PMID 12583960
- [Background] Mazzaferri EL. An overview of the management of papillary and follicular thyroid carcinoma. Thyroid. 1999 May;9(5):421-7. doi: 10.1089/thy.1999.9.421. PMID 10365671
- [Background] Mazzaferri EL, Jhiang SM. Long-term impact of initial surgical and medical therapy on papillary and follicular thyroid cancer. Am J Med. 1994 Nov;97(5):418-28. doi: 10.1016/0002-9343(94)90321-2. PMID 7977430
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-DK-0025.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 87 patients were screened for the eligibility for this study. Total of 34 patients were enrolled into the study
Pre-assignment Details: The sample size for the trial is 100 patients and the goal for the number of patients to be randomized by November 2010 is 74 patients.
Period: Overall Study
Arm/Group | Lithium Carbonate | Placebo
Started | 17 | 17
Completed | 15 | 14
Not Completed | 2 | 3
Not completed — Physician Decision | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lithium Carbonate | Placebo | Total
Number analyzed (Participants) | 15 | 14 | 29
Age Continuous [Mean (Standard Deviation); unit: years] | 39.8 (11.8) | 38.6 (10.2) | 39.2 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 3 | 2 | 5
Race/Ethnicity, Customized [Number; unit: Participants]
  African American | 1 | 1 | 2
  Caucasian | 12 | 13 | 25
  Hispanic | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Successful Thyroid Ablation as Defined by Negative Recombinant Human Thyrotropin (rhTSH) Stimulated Radioiodine Whole Body Scan (RAI WBS) at 1 Year.
Time Frame: 1 year
Measure: Number; unit: Participants
Arm/Group | Lithium Carbonate | Placebo
Number analyzed (Participants) | 15 | 14
Participants | 10 | 10

ADVERSE EVENTS:
Arm/Group | Lithium Carbonate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium Carbonate (N=15) | Placebo (N=14)
Acute respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes